CLINICAL TRIAL: NCT05889026
Title: The Effect of Extracorporeal Shock Wave Therapy After Botulinum Toxin Type A Injection for Post-stroke Spasticity: Preliminary Study, Randomized Controlled Trials
Brief Title: The Effect of Extracorporeal Shock Wave Therapy After Botulinum Toxin Type A Injection for Post-stroke Spasticity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESWT RCT
Record Dates: First submitted 2023-05-09; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Stroke; Hemiplegia, Spastic; Muscle Spasticity
MeSH Terms: conditions — Stroke; Hemiplegia; Muscle Spasticity | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botulinum toxin treatment with extracorporeal shock wave therapy (Active Comparator): Nabota® (Daewoong Pharmaceutical Co. Ltd., Seoul, Korea) was used. It was diluted with 0.9% sodium chloride solution and injected into the bellies of the upper-extremity muscles.
  ESWT was performed immediately after botulinum toxin injection and was performed once a day for 5 days. Three weeks and 3 months after ESWT, spasticity was evaluated.
  Interventions: Device: Extracorporeal shock wave therapy; Procedure: Botulinum toxin treatment
- Botulinum toxin treatment only (Sham Comparator): Nabota® (Daewoong Pharmaceutical Co. Ltd., Seoul, Korea) was used. It was diluted with 0.9% sodium chloride solution and injected into the bellies of the upper-extremity muscles. Three weeks and 3 months after Botox treatment, spasticity was evaluated.
  Interventions: Procedure: Botulinum toxin treatment

INTERVENTIONS:
Device: Extracorporeal shock wave therapy — Stimulation was given to the brachial muscle, 1000 times, 4Hz, and energy flux density was 0.030mJ/mm2.
  Arms: Botulinum toxin treatment with extracorporeal shock wave therapy
Procedure: Botulinum toxin treatment — The toxin dose was established for each patient: it ranged between 80 unit and 300 unit.

SUMMARY:
There are few studies on whether botulinum toxin treatment and extracorporeal shock wave therapy are more effective than botulinum toxin alone treatment for post-stroke spasticity.

DETAILED DESCRIPTION:
If the study results can be drawn that the group receiving extracorporeal shock wave therapy along with botulinum toxin treatment can increase the effect of botulinum toxin treatment and lengthen the treatment period compared to the group with botulinum toxin treatment only, it can be widely used as an auxiliary treatment for botulinum toxin treatment. This study was carried out with the expectation that it would be possible to provide a basis for this.

ELIGIBILITY:
Inclusion Criteria:

1. at least 6 weeks after stroke diagnosis
2. upper-extremity (elbow, wrist and finger) spasticity Modified Ashworth Scale (MAS) score > 2
3. ability to stand and walk safely without help or assistance

Exclusion Criteria:

1. improper indication for botulinum toxin A (BTxA) injection, for example, myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, and motor neuropathy
2. previous contracture and/or deformity of the upper extremities
3. concurrent peripheral neuropathy and/or myopathy
4. difficulty in participating in the study due to cognitive impairment.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-09-08 (Actual)

PRIMARY OUTCOMES:
Modified ashworth scale of upper extremities spasticity | Pre-treatment (baseline)
  minimum grade 0, maximum grade 4 / higher grade means severe spasticity
Modified ashworth scale of upper extremities spasticity | Three weeks after treatment
  minimum grade 0, maximum grade 4 / higher grade means severe spasticity
Modified ashworth scale of upper extremities spasticity | Three months after treatment
  minimum grade 0, maximum grade 4 / higher grade means severe spasticity

SECONDARY OUTCOMES:
Modified tardieu scale of upper extremities spasticity | Pre-treatment (baseline)
  Unit : degree / higher degree means little limitation of range of motion
Modified tardieu scale of upper extremities spasticity | Three weeks after treatment
  Unit : degree / higher degree means little limitation of range of motion
Modified tardieu scale of upper extremities spasticity | Three months after treatment
  Unit : degree / higher degree means little limitation of range of motion
Fugl-Meyer assessment of upper extremity Fugl-Meyer assessment of upper extremity Fugl-Meyer assessment of upper extremity Fugl-Meyer assessment of upper extremity | Pre-treatment (baseline)
  Minimum score 0, maximum score 66 / higher score means better function of upper extremity
Fugl-Meyer assessment of upper extremity | Three months after treatment
  Minimum score 0, maximum score 66 / higher score means better function of upper extremity
Action research arm test | Pre-treatment (baseline)
  Minimum score 0, maximum score 57 / higher score means better function of upper extremity
Action research arm test | Three weeks after treatment
  Minimum score 0, maximum score 57 / higher score means better function of upper extremity
Action research arm test | Three months after treatment
  Minimum score 0, maximum score 57 / higher score means better function of upper extremity
Modified barthel index | Pre-treatment (baseline)
  Minimum score 0, maximum score 100 (if w/c ambulation, 90) / higher score means better capacity for activities of daily living
Modified barthel index | Three weeks after treatment
  Minimum score 0, maximum score 100 (if w/c ambulation, 90) / higher score means better capacity for activities of daily living
Modified barthel index | Three months after treatment
  Minimum score 0, maximum score 100 (if w/c ambulation, 90) / higher score means better capacity for activities of daily living

CONTACTS AND LOCATIONS:
Locations (1):
- Korea university guro hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No